CLINICAL TRIAL: NCT02975440
Title: Non-randomized, Non-blinded, Non-placebo-controlled Study to Investigate the Influence of Repeated Daily Administration of 600 mg Rifampicin Given Once Daily Over 11 Days on the Pharmacokinetics, Safety, and Tolerability of a Single Oral Dose of 4 mg Vilaprisan in Healthy Postmenopausal Women.
Brief Title: Drug-drug Interaction Study Between Orally Administered Rifampicin and Vilaprisan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17773
Record Dates: First submitted 2016-11-04; First posted 2016-11-29 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Endometriosis
Keywords: Vilaprisan; PK; rifampicin; midazolam,; CYP3A4 induction; drug-drug interaction
MeSH Terms: conditions — Endometriosis | interventions — Rifampin; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Treatment A (Period 1): a single oral dose of 4 mg Vilaprisan and 1 mg Midazolam Treatment B (Period 2): 600 mg Rifampicin once daily (qd) for 7 days followed by administration of a single oral dose of 4 mg Vilaprisan and 1 mg Midazolam followed by 600 mg Rifampicin 12 hours after Vilaprisan and Midazolam administration and continued dosing of 600 mg Rifampicin once daily for 3 days
  Interventions: Drug: Rifampicin; Drug: Midazolam; Drug: BAY1002670_Vilaprisan

INTERVENTIONS:
Drug: Rifampicin — 11 single oral doses of 600 mg Rifampicin resulting in a total dose of 6600 mg Rifampicin.
Drug: Midazolam — 2 single oral doses of 1 mg Midazolam resulting in a total dose of 2 mg Midazolam
Drug: BAY1002670_Vilaprisan — 2 single oral doses of 4 mg Vilaprisan resulting in a total dose of 8 mg Vilaprisan

SUMMARY:
This study will be conducted in a single center, open-label study with a single group fixed sequence design to evaluate the effect of repeated oral administration of 600 mg RIF(Rifampicin) given once daily over 11 days on the single oral dose pharmacokinetics of VPR(Vilaprisan) and on MDZ(Midazolam) as a reference (probe) substance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female postmenopausal subjects
* Age: 45 to 65 years (inclusive)
* Body mass index (BMI) : ≥20 and ≤32 kg/m²
* Race: White

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Relevant diseases within the last 4 weeks prior to the first drug administration
* Existing chronic diseases requiring medication
* Known or suspected malignant tumors (including history of malignant tumors, with a status after treatment), known or suspected benign tumors of the liver and pituitary (including after treatment)
* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Regular use of medicines
* Repeated use of drugs during 1 week before first study drug administration which might affect absorption (e.g. laxatives, loperamide, metoclopramide, antacids, H2-receptor antagonists)

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-04-11 (Actual)

PRIMARY OUTCOMES:
AUC of Vilaprisan in plasma with co-medication Rifampicin | blood sampling for pharmacokinetics of Vilaprisan (LC-MS/MS) at the following time points post administration of Vilaprisan and Midazolam: 0.5,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,15 hour, thereafter daily sampling up to 14 days
Cmax of Vilaprisan in plasma with co-medication Rifampicin | blood sampling for pharmacokinetics of Vilaprisan (LC-MS/MS) at the following time points post administration of Vilaprisan and Midazolam: 0.5,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,15 hour, thereafter daily sampling up to 14 days
AUC of Vilaprisan in plasma without co-medication Rifampicin | blood sampling for pharmacokinetics of Vilaprisan (LC-MS/MS) at the following time points post administration of Vilaprisan and Midazolam: 0.5,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,15 hour, thereafter daily sampling up to 14 days
Cmax of Vilaprisan in plasma without co-medication Rifampicin | blood sampling for pharmacokinetics of Vilaprisan (LC-MS/MS) at the following time points post administration of Vilaprisan and Midazolam: 0.5,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,15 hour, thereafter daily sampling up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, Germany